CLINICAL TRIAL: NCT00851292
Title: The BIOPRES Trial; Transrectal BIOpsies of the PRostate: End Versus Side-firing
Brief Title: The BIOPRES Trial: Transrectal BIOpsies of the PRostate: End Versus Side-firing
Acronym: BIOPRES
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amphia Hospital (Other)
Responsible Party: S. Roemeling, Amphia hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: ROE-3
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; biopsy; TRUS; diagnosis
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Side-firing (Active Comparator): prostate biopsies obtained with side-firing probe
  Interventions: Device: TRUS probe
- End-firing (Active Comparator)
  Interventions: Device: TRUS probe

INTERVENTIONS:
Device: TRUS probe — end-firing and side-firing vary in the angle in which they sample the prostate

SUMMARY:
The purpose of this study is to study the difference in prostate cancer between two prostate biopsy techniques, namely end-firing and side-firing. These differ in the angle at which the prostate is biopsied.

DETAILED DESCRIPTION:
Rationale: Research towards the efficacy of transrectal prostate biopsies has predominantly focused on the amount of biopsy cores. However, variation in the angle of entrance of the biopsy gun has been less studied. It is believed that obtaining biopsy cores by end firing will improve the efficacy, because of an improved sampling of the apical region.

Objectives: To investigate the difference between side and end-firing in transrectal prostate needle biopsies in terms of qualitative and quantitative prostate cancer detection.

Methods: From September 1st 2009 - September 1st 2012, all men with an initial prostate biopsy in a representative, Dutch, general hospital with six participating urologists and two residents will be subjected to a randomized controlled, single blind, single center, diagnostics trial. Men will be randomized for a biopsy using an end-firing or a side-firing probe. The primary endpoint is the prostate cancer detection rate; secondary endpoints are the number of cores invaded with prostate cancer, nomogram for indolent cancer-score, Gleason score, complications and biopsy length.

Expected outcomes: We hypothesize that no differences between the biopsy techniques exist.

ELIGIBILITY:
Inclusion Criteria:

* PSA and DRE performed in advance of the biopsy
* Informed consent
* Number of biopsy cores according to the volume dependent biopsy protocol (8 cores in prostates with a volume less than 40 mL., 10 in 40-60 mL. and 12 in >60 mL.)

Exclusion Criteria:

* None

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2009-10; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
The presence of prostate cancer in the tissue obtained by prostate needle biopsy | This outcome parameter will be available 5 days after the biopsy has been done. E.g. there will be virtually no 'follow-up' period.

SECONDARY OUTCOMES:
Number of cores invaded with prostate cancer | All secondary outcome measures, except for the complications will be available when the pathology report emerges. Initial complications will be registered after 2 weeks.
Gleason score | All secondary outcome measures, except for the complications will be available when the pathology report emerges. Initial complications will be registered after 2 weeks.
Complications | All secondary outcome measures, except for the complications will be available when the pathology report emerges. Initial complications will be registered after 2 weeks.
Biopsy length | All secondary outcome measures, except for the complications will be available when the pathology report emerges. Initial complications will be registered after 2 weeks.
Nomogram score for indolent prostate cancer | All secondary outcome measures, except for the complications will be available when the pathology report emerges. Initial complications will be registered after 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Stijn Roemeling, MD, PhD, Principal Investigator — Amphia Hospital
Locations (1):
- Amphia hospital, Breda, North Brabant, Netherlands